CLINICAL TRIAL: NCT06174415
Title: An Exploratory Study of Visual Function Rehabilitation in Patients With Ocular Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023KYPJ122
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-05

CONDITIONS: Eye Injuries
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Intervention Model Description: Comparing the data before and after treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The experimental group consisted of the patients themselves. Compare data before and after treatment
  Interventions: Device: Perceptual Learning

INTERVENTIONS:
Device: Perceptual Learning — Perceptual training is carried out at home once a day, and the viewing distance of the patients from the display screen is uniformly 1.5m, 30 minutes each time, for three months, and they return to the hospital for re-examination of ophthalmology at the 3rd months after the training. When using the perceptual training program for the first time, the training program will adjust the size of the Gabor spot according to the size of the user's computer, and prompt the patient to adjust the brightness of the computer screen to unify the Gabor spot parameters of each user and ensure the consistency of the spot stimulation information received by each user.

SUMMARY:
Ocular trauma is one of the leading causes of blindness worldwide, often resulting in severe visual impairment or even loss of vision after injury.

Although after powerful surgical treatment, there are still some patients whose visual function is difficult to improve, and the patients with eye trauma lack effective vision rehabilitation therapy.Therefore, the research on visual function rehabilitation of patients with ocular trauma needs to be further carried out . Perceptual learning is based on cortical remodeling, repetitive visual task training. This training is to perform a series of repetitive visual tasks through the Gabor patch, simulating the receptive field structure of simple cells in the primary visual cortex (V1 area), "awakening visual cells", and improving the visual processing ability of the cerebral cortex. Compared with the traditional vision rehabilitation therapy, perceptual learning optimizes the visual quality at the visual center level. It is an innovative therapy, having the potential to solve the visual function of patients with eye trauma. This study intends to explore new visual rehabilitation methods for patients with ocular trauma, and explore the changes in visual cortical function and area of patients after perceptual training.

DETAILED DESCRIPTION:
Perceptual training is a type of perceptual learning that initiates neural modifications during continuous repetitive task training, thereby increasing neural efficiency and improving the visual processing capabilities of the cerebral cortex. The perceptual training program simulates the receptive field structure of simple cells in the primary visual cortex (area V1) through Gabor cursors and lateral occlusion techniques to awaken visual cells during repetitive visual tasks. Gabor Patches are targeted stimuli that are widely used in the field of optic neurology to produce highly effective stimulation of the primary visual cortex. Lateral shading technology can effectively stimulate specific neurons. It can not only improve the interaction of neurons in the cerebral cortex in patients with amblyopia, but also stimulate the cooperation of neurons. This technology has also been proved to be effective in normal people. Therefore, on the basis of this theory, we plan to use perceptual learning to conduct repetitive visual stimulation for three months, and return to visit three times within three months. The main indicator is contrast sensitivity, and the efficacy of perceptual learning is evaluated by evaluating the improvement of contrast sensitivity. The study was designed as a self-controlled before-and-after trial. Volunteers were recruited from the outpatients of Zhongshan Ophthalmic Center's ophthalmic trauma clinic to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Retinopathy, optic neuropathy, endophthalmitis and other injuries caused by ocular trauma, with varying degrees of central vision reduction and visual field impairment
2. Age 3~60 years old
3. Best corrected visual acuity of the affected eye: 20/200≤BCVA≤20/25
4. Intraocular pressure is normal, non-hypotonal/atrophic: 7--21mmHg
5. After the traumatic injury, the condition is stable ≥for 3 months after treatment, and the visual axis has a complete and transparent optical pathway
6. If the patient is injured in one eye, There were no abnormal lesions in the contralateral eye, no abnormalities in slit lamp and indirect ophthalmoscopy, and no peripheral retinopathy in both eyes was found on triprimmoscopy. Carefully ask for a history of no other eye disease in both eyes and a systemic history that has caused an associated eye disease or has affected visual formation.
7. The cranial structure is intact, the function is good, and there is no primary or secondary injury
8. Able to cooperate with the questionnaire and treatment, good compliance
9. Those who are willing to sign the informed consent form

Exclusion Criteria:

1. Have active inflammation of the eye
2. Previous abnormal intraocular blood supply such as occlusion of the central intraocular artery due to trauma or non-traumatic factors
3. History of other non-traumatic intraocular surgery
4. Ocular related lesions caused by other non-traumatic factors that can interfere with this study, such as age-related macular degeneration, glaucoma, amblyopia, etc.
5. Use of other rehabilitation training methods or visual aids 3 months before enrollment
6. Lesions with systemic diseases whose degree of lesions have affected visual function, such as diabetic retinopathy, Hypertension and arteriosclerotic fundus changes, rubella-related ocular changes, etc.
7. Patients with severe systemic diseases such as renal failure and malignant hypertension or may affect visual function (such as retinal structure and function, choroidal structure and function, etc.)
8. Patients with congenital ocular lesions
9. Patients with optic nerve and retinopathy caused by non-traumatic factors
10. Patients with cranial brain disease or craniocere-related lesions with poor cortical function
11. Psychological related diseases
12. MRI contraindications, Such as claustrophobia and non-MRI compatible metal implants
13. people with speech impairment and intellectual disability
14. those who are considered inappropriate by the investigator

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 3 months
  Log MAR

SECONDARY OUTCOMES:
Contrast Sensitivity Function | 3 months
  Area Under the Log Contrast Sensitivity Function

CONTACTS AND LOCATIONS:
Overall Officials: XUEYING ZHONGLIU, Study Director — Zhonshan Ophthalmic Center, Sun-Yat-sen University Organization
Locations (1):
- Zhonshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided